CLINICAL TRIAL: NCT05609825
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3875383 in Healthy Participants and Participants With Hypertriglyceridemia
Brief Title: A Study of LY3875383 in Healthy Participants and Participants With Hypertriglyceridemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in risk/benefit ratio, which no longer favoured continued development.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18537; J4D-MC-EZFA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-04; First posted 2022-11-08 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LY3875383 (Part A) (Experimental): Single-ascending doses of LY3875383 administered subcutaneously (SC).
  Interventions: Drug: LY3875383
- LY3875383 (Part B) (Experimental): Single doses of LY3875383 administered SC.
  Interventions: Drug: LY3875383
- LY3875383 (Part C) (Experimental): Single doses of LY3875383 administered SC.
  Interventions: Drug: LY3875383
- LY3875383 (Part D) (Experimental): Single doses of LY3875383 administered SC.
  Interventions: Drug: LY3875383
- Placebo (Part A) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part C) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Placebo (Part D) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3875383 — Administered SC.
  Arms: LY3875383 (Part A); LY3875383 (Part B); LY3875383 (Part C); LY3875383 (Part D)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C); Placebo (Part D)

SUMMARY:
The main purpose of this study is to determine the tolerability and side effects related to LY3875383 given as a single injection under the skin to healthy participants and participants with elevated triglyceride (TG) levels.The study will also assess how fast LY3875383 gets into the blood stream and how long the body takes to get rid of it. Each enrolled participant will receive a single dose of either LY3875383 or placebo.The study will be conducted in four parts (A, B, C and D) and may last up to approximately 28 to 56 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Have a body mass index (BMI) between 18.5 and 40 kilograms per square meter (kg/m²), inclusive.
* Males who agree to follow contraceptive requirements, or women not of childbearing potential (WNOCBP).

Healthy participants (Part A):

• Participants must be overtly healthy, as determined by medical evaluation.

For Part B:

• Participants must be first-generation Japanese, defined as the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan.

Hypertriglyceridemia participants (Parts C and D):

For Part C:

* Have history of very high triglyceride (lipid) level 500 mg/dL ≤ TG <2000 mg/dL, which needs to be further confirmed at screening.
* Participants must be on a lipid-modifying diet and can be on stable lipid-lowering drugs (LLDs) for at least 8 weeks before screening and plan to continue the same throughout the study duration.

For Part D:

* Have history of high triglyceride (lipid) level between 150 mg/dL and 500 mg/dL inclusive at pre-screening or based on medical history and confirmed at screening and Low-density lipoprotein cholesterol (LDL-C) level of ≥40 mg/dL.
* Participants must be on a stable moderate or high-intensity dose of a statin for at least 8 weeks before screening and plan to continue the same medication and dose throughout the study duration.

Exclusion Criteria:

All participants:

* Participants must not be currently participating in or completed a clinical trial within the last 30 days
* Have donated blood of more than 500 mL within the previous 3 months
* Have one of the following viral infections: hepatitis B virus, hepatitis C virus or human immunodeficiency virus (HIV).
* Participants must not be heavy alcohol drinkers or cigarette smokers.

For Part C: Have active pancreatitis within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 53
  A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK):Area Under the Concentration Versus Time Curve (AUC) of LY3875383 | Predose up to Day 8 post dose
  PK: AUC of LY3875383
PK: Maximum Observed Concentration (Cmax) of LY3875383 | Predose up to Day 8 post dose
  PK: Cmax of LY3875383
Part C and D only: Pharmacodynamics (PD): Percentage Change from Baseline in Fasting Triglyceride (TG) | Baseline through up to Week 53
  Part C and D only: PD: Percentage Change from Baseline in Fasting TG
Part D only: PD: Percentage Change from Baseline in Fasting Non-High-Density Lipoprotein Cholesterol (HDL-C) | Baseline through Week 53
  Part D only: PD: Percentage Change from Baseline in Fasting non-HDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3875383 in Healthy Participants and Participants With Hypertriglyceridemia — https://trials.lilly.com/en-US/trial/366875